CLINICAL TRIAL: NCT04883814
Title: 18F-fluoroestradiol (FES) PET/CT Compared To Standard-of-Care Imaging In Patients With Breast Cancer
Brief Title: 18F-fluoroestradiol (FES) PET/CT for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Gary Ulaner, Director Molecular Imaging and Therapy, Hoag Memorial Hospital Presbyterian
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 182-20-CA
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: 18F-fluoroestradiol; Breast Cancer; PET/CT; Staging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Initial Staging (Experimental): FES PET/CT will be compared to CT/bone scan for detection of unsuspected distant metastases in patients with ER-positive locally advanced breast cancer
  Interventions: Diagnostic Test: 18F-fluoroestradiol PET/CT
- Suspected disease recurrence (Experimental): FES PET/CT will be compared to CT/bone scan for detection of unsuspected distant metastases in patients with ER-positive breast cancer and suspected disease recurrence
  Interventions: Diagnostic Test: 18F-fluoroestradiol PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-fluoroestradiol PET/CT — Estrogen receptor targeted imaging
  Other Names: FES PET/CT

SUMMARY:
The standard of care imaging of breast cancer metastases recommended by the National Comprehensive Cancer Network (NCCN), CT of the chest/abdomen/pelvis and bone scan, may be suboptimal. 18F-fluoroestradiol (FES) is a novel PET tracer designed to detect estrogen receptors, which are often expressed in breast cancers. FES PET/CT may provide improved evaluation of metastases in patients with ER-positive breast cancer.

DETAILED DESCRIPTION:
This will be a phase II clinical trial to assess the clinical value of FES for staging and detection of disease recurrence in patients with ER-positive breast cancer, in direct comparison to the National Comprehensive Cancer Network's (NCCN) recommended standard-of-care using CT of the chest/abdomen/pelvis and bone scan [2].

Two cohorts will be evaluated:

1. Patients with advanced local breast cancer that will undergo standard of care imaging (CT + bone scan) to evaluate for unsuspected distant metastases.
2. Patients with suspicion for breast cancer recurrence that will undergo standard of care imaging (CT + bone scan) to evaluate for disease recurrence.

In both cohorts, FES PET/CT will be obtained, and compared with standard of care imaging. Whether on standard of care imaging or the research FES PET/CT, lesions suspicious for unsuspected distant metastases (cohort 1) or the site of disease recurrence (cohort 2) will be selected for biopsy, as is clinically standard of care to confirm disease that would alter patient management. Pathology will be used as the reference standard for confirming malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 years of age.
2. Histologically confirmed ER-positve breast cancer. Any pathology from a primary or metastatic breast cancer site demonstrating ER-positivity will be allowed.
3. ECOG performance status 0 to 2
4. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
5. Either:

   1. For cohort 1: Stage 2B-3C locally advanced disease and plan for CT/bone scan systemic staging or
   2. For cohort 2: Suspected recurrent disease and plan for CT/bone scan systemic staging

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Patients who cannot undergo PET/CT scanning because of weight limits. PET/CT scanners may not be able to function with patients over 450 pounds.
4. Selective ER Modulators (SERMs) such as tamoxifen and Selective ER Degraders (SERDs) such as fulvestrant may reduce detection of ER-positive lesions by FES. Thus, exclusion criteria specify that patients must be withdrawn from Selective ER Modifiers for at least 8 weeks and withdrawn from Selective ER Degraders for for least 24 weeks prior to performance of the FES PET/CT.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Detection of unsuspected distant metastases | up to 4 weeks
  FES PET/CT will be compared against standard of care CT/bone scan for detection of unsuspected distant metastases in patients with ER+ locally advanced disease

SECONDARY OUTCOMES:
Detection of suspected disease recurrence | up to 4 weeks
  FES PET/CT will be compared against standard of care CT/bone scan for detection of unsuspected distant metastases in patients with ER+ breast cancer and suspected disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ulaner, MD, PhD, Principal Investigator — Hoag Family Cancer Institute
Locations (1):
- Hoag Memorial Hospital Presbyterian, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller R, Battle M, Wangerin K, Huff DT, Weisman AJ, Chen S, Perk TG, Ulaner GA. Evaluating Automated Tools for Lesion Detection on 18F Fluoroestradiol PET/CT Images and Assessment of Concordance with Standard-of-Care Imaging in Metastatic Breast Cancer. Radiol Imaging Cancer. 2025 May;7(3):e240253. doi: 10.1148/rycan.240253. PMID 40314583
- [Derived] Ulaner GA, Silverstein M, Nangia C, Tetef M, Vandermolen L, Coleman C, Khan S, MacDonald H, Patel T, Techasith T, Mauguen A. ER-Targeted PET for Initial Staging and Suspected Recurrence in ER-Positive Breast Cancer. JAMA Netw Open. 2024 Jul 1;7(7):e2423435. doi: 10.1001/jamanetworkopen.2024.23435. PMID 39058489